CLINICAL TRIAL: NCT00004833
Title: Randomized Study of Plasmapheresis or Human Immunoglobulin Infusion in Childhood Guillain-Barre Syndrome
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Organization: FDA Office of Orphan Products Development (U.S. Federal Agency)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: 199/13444; EUSM-076-97; EUSM-FDR001265
Record Dates: First submitted 2000-02-24; First posted 2000-02-25 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2002-09

CONDITIONS: Guillain-Barre Syndrome
Keywords: Guillain-Barre syndrome; demyelinating neuropathy; neurologic and psychiatric disorders; rare disease
MeSH Terms: conditions — Guillain-Barre Syndrome; Neurologic Manifestations; Mental Disorders; Rare Diseases | interventions — Immunoglobulins

INTERVENTIONS:
Drug: Immune globulin

SUMMARY:
OBJECTIVES:

I. Compare the efficacy of plasmapheresis and human immunoglobulin infusion in minimizing morbidity and augmenting the pace of recovery in children with Guillain-Barre syndrome.

II. Compare the potential risks, in terms of treatment related side effects and adverse clinical outcome, between these two treatment modalities.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE:

This is a randomized, multicenter study.

Patients are randomized to receive either human immunoglobulin infusion (IVIg) (arm I) or plasmapheresis (arm II).

Arm I patients receive liquid heat-treated IVIg for 4 days starting on day 1 and then another single infusion of IVIg on day 7, 8, or 9.

Arm II patients receive serial plasmapheresis treatments. The first exchange is given on day 1 and the remaining exchanges are given over the next 5-10 days.

Patients are followed at weeks 1, 2, 3, 4, 8, 12, and 24.

Completion date provided represents the completion date of the grant per OOPD records

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

Guillain-Barre syndrome (GBS): Progressive weakness of two or more limbs; Absence or reduced tendon reflexes; No atypical symptoms of GBS (e.g., Miller-Fisher variant); No pure sensory neuropathy; No prior history of GBS

Disability at least grade 3 according to Guillain-Barre Study Group grading scale (unable to walk 5 meters without assistance); Must not have improvement of one or more disability grades prior to randomization in this study

No paresthesias, numbness, or weakness that began more than 14 days before randomization in this study

No CNS involvement

--Prior/Concurrent Therapy--

Biologic therapy: No prior treatment with plasmapheresis or infusion of human immunoglobulin (IVIg)

Endocrine therapy: No concurrent corticosteroids or other immunosuppressants (except for concurrent medical conditions, e.g., asthma)

Radiotherapy: Not specified

Surgery: Not specified

Other: No concurrent mechanical ventilation

--Patient Characteristics--

Age: Under 18 but with at least 3 months of independent walking

Hematopoietic: Cerebrospinal fluid leukocyte count less than 50/mm3

Hepatic: No liver failure

Renal: No kidney failure

Neurological: No other major neurologic diseases, other neuromuscular disorders, or cerebral palsy

Other: HIV negative; No contraindications to plasmapheresis or IVIg; No severe uncontrolled infection; No known IgA hypersensitivity; No other preexisting disease that would interfere with assessment of disability grades; No other causes of acquired weakness (e.g., poliomyelitis, botulism, or other etiologies); No diabetes; Not pregnant

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 170
Dates: Start 1995-07; Study Completion 2002-11

CONTACTS AND LOCATIONS:
Overall Officials: John T. Sladky, Study Chair — Emory University